CLINICAL TRIAL: NCT01217242
Title: Cross-sectional Descriptive Study to Quantify to What Extent Activity Capacity, Performance and Body Composition Predict Day to Day Life Participation in Ambulatory Children With CP.
Brief Title: Activity and Participation in Ambulatory Cerebral Palsy
Acronym: APCP
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kristie Bjornson, Assistant Professor Pediatrics, Seattle Children's Hospital
Other Study IDs: K23HD060764 (NIH); K23HD060764 (NIH)
Record Dates: First submitted 2010-10-04; First posted 2010-10-08 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; walking activity; physical activity; participation; activity performance; activity capacity
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with cerebral palsy (CP): ages 2 to < 10 years who are able to walk with or without an assistive device

SUMMARY:
The investigators would like to understand how the physical activity levels and body size of a child with cerebral palsy (CP) in a clinical situations versus out in the community relates to what they want to do in day to day life (participation in life). The investigators believe that what a child really does out in day to day life will predict life participation to a greater degree than what they do in a structured clinical situation (i.e. therapy session with therapist). The investigators think that increased body size with normal growth is related to less physical activity and participation in day to day life for children with cerebral palsy (CP) who can walk. This project will use a novel accelerometer to measure walking activity during day to day life.

DETAILED DESCRIPTION:
We want to know how the physical activity of children with walking problems or cerebral palsy (CP) relates to what they do in their day to day lives.

We are looking for children who:

* Have walking problems that started before age 2
* Have any type of cerebral palsy (CP) or primary problem that is a developmental movement disorder
* May have hemiplegia, diplegia, walking quadriplegia, May have ataxia, spastic, mixed tone, athetoid, or dyskinetic
* Ages 2 years to less than 10 years
* Able to do some functional walking with or without help(walkers, gait trainers)
* Project requires a one time visit to Seattle Children's Hospital of about 2 hours.
* Children and/or parents will complete surveys.
* The child will be tested for their gross motor and walking skills like at a physical therapy session.
* The child will be given an ankle monitor to wear for 7-10 days.
* They will return the monitor by mail with a questionnaire about what they did the last week.
* Families will receive a print out of their child's walking activity

ELIGIBILITY:
Inclusion Criteria:

1. age 2 to <10 years (30 per four age groups/2 year increments)
2. Gross Motor Function Classification System (GMFCS) levels I-III
3. diagnosis of cerebral palsy (CP) or developmental movement disorder that occurred prior to age two.

Exclusion Criteria:

1. visual impairment limiting physical activity
2. lower extremity botox injections in the last 3 months
3. uncontrolled seizure disorder impacting mobility skills
4. orthopedic or neurosurgery in the last 6 months.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy (CP) or developmental movement disorder before age two who are able to walk
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Community walking activity with the STEPWATCH accelerometer | Assessed at one time point with a 7-10 walking sample
  Walking activity performance within the context of daily life will be measured with a monitor called the StepWatch. The StepWatch was specifically designed and validated for long-term assessment of ambulatory activity during day-to-day life. It is a small,waterproof, self-contained device that is worn on the ankle. It records the number of strides taken every minute for up to two months between downloads.

SECONDARY OUTCOMES:
Participation in day to day life activities | Assessed as one time point by parental/child report of participation in the last 4 months
  Participation will be quantified by two valid measures of pediatric life participation, the Children's Assessment of Participation and Enjoyment (CAPE) and the Assessment of Life Habits (Life-H for Children).The CAPE was designed to document the child's report of participation in day to day activities, while the Life-H for children is intended to describe a group of life habits that are characteristic of children in their environment (home, school and neighborhood).

CONTACTS AND LOCATIONS:
Overall Officials: Carol Nicholson, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States